CLINICAL TRIAL: NCT01063816
Title: A Phase 1 Study of Veliparib in Combination With Carboplatin and Gemcitabine in Subjects With Advanced Solid Tumors
Brief Title: A Study of ABT-888 in Combination With Carboplatin and Gemcitabine in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10-758
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Advanced Solid Tumors
Keywords: PARP Inhibitors
MeSH Terms: interventions — veliparib; Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: veliparib (ABT-888); Drug: carboplatin; Drug: gemcitabine

INTERVENTIONS:
Drug: veliparib (ABT-888) — Dosing orally twice daily starting Cycle 2 Day 1- through 21 adjusted for subsequent cohorts using a continuous reassessment method.
Drug: carboplatin — Carboplatin will be dosed on Day 1 of each cycle, intravenously.
Drug: gemcitabine — Dosing on Days 1 and 8 of each Cycle, intravenously.
  Other Names: Gemzar

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose of veliparib (ABT-888)and to establish the recommended Phase 2 dose of veliparib (ABT-888) when administered in combination with carboplatin and gemcitabine in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid tumors that are metastatic or unrespectable for which carboplatin/gemcitabine is a treatment option.
* Eastern Cooperative Group performance score of 0 to 2.
* Adequate hematologic, hepatic and renal function
* Subject has received up to 2 DNA damaging or cytotoxic regimens in the past five years

Exclusion Criteria:

* Subject has received any anti-cancer therapy including chemotherapy, immunotherapy, radiotherapy, biologic or any investigational therapy within 28 days prior to study administration.
* Subjects with known history of brain metastases and primary CNS tumors.
* Hypersensitivity reactions to platinum compounds or gemcitabine.
* Clinically significant and uncontrolled major medical conditions
* Active malignancy within the past 5 years except for any cancer in situ cured or non-melanoma carcinoma of the skin.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2010-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose and recommended Phase 2 dose | ABT-888 will be dose escalated until the largest dose is reached based on the probability of dose, limiting toxicities is based per continual reassessment method (CRM).

SECONDARY OUTCOMES:
Pharmacokinetics Area Under the Curve (AUC) | Timepoints: 30 and 45 minutes, 1,1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5,6,6.5, 7 and 8 hours past dose
Safety assessment: Electrocardiogram | Screening, Day 8 of each Cycle of drug and Final Visit
Safety assessment: Clinical Laboratory Tests | Screening, Day 1 and Day 8 of each cycle, Final Visit and 30 Day Follow-up Visit
  Hematology and Chemistry
Physical exam including vital signs | Screening, Cycle 1 Day 8, Day 1 of all cycles starting with Cycle2, Final Visit and 30 Day Follow-up Visit
  Physical exam including blood pressure, pulse and temperature
Safety assessment: Adverse event assessments | All study visits
  Collect all adverse events at each visit
Tumor assessment | Screening, every nine weeks and Final Visit
  Computerized tomography (CT) scan of chest, abdomen and pelvis to assess tumor burden

CONTACTS AND LOCATIONS:
Overall Officials: Mark D McKee, MD, Study Director — AbbVie

REFERENCES:
- [Background] Gray HJ, Bell-McGuinn K, Fleming GF, Cristea M, Xiong H, Sullivan D, Luo Y, McKee MD, Munasinghe W, Martin LP. Phase I combination study of the PARP inhibitor veliparib plus carboplatin and gemcitabine in patients with advanced ovarian cancer and other solid malignancies. Gynecol Oncol. 2018 Mar;148(3):507-514. doi: 10.1016/j.ygyno.2017.12.029. Epub 2018 Jan 17. PMID 29352572
- See also: Related Info — https://doi.org/10.1016/j.ygyno.2014.03.151